CLINICAL TRIAL: NCT01009970
Title: Multicenter Study of Phase II With Rituximab, Cyclophosphamide, Doxorubicin Liposomal (Myocet ®), Vincristine, Prednisone, (R-COMP) in Non-Hodgkin's Lymphoma Diffuse Large B Cell in Cardiopathic Patients
Brief Title: Study With Rituximab, Cyclophosphamide, Doxorubicin Liposomal (Myocet®), Vincristine, Prednisone, (R-COMP) to Treat Non-Hodgkin's Lymphoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fondazione Italiana Linfomi - ETS (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIL-HEART01; 2009-012143-42
Record Dates: First submitted 2009-11-06; First posted 2009-11-09 (Estimated); Last update posted 2011-10-13 (Estimated); Status verified 2011-10

CONDITIONS: Diffuse Large B-Cell Lymphoma
Keywords: Diffuse Large B-Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — Rituximab; Cyclophosphamide; Vincristine; Prednisone; Doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): R-COMP
  Interventions: Drug: Rituximab; Drug: Cyclophosphamide; Drug: Vincristine; Drug: Prednisone; Drug: Doxorubicin

INTERVENTIONS:
Drug: Rituximab — 375 mg/m2 day 1
Drug: Cyclophosphamide — 750 mg/m2 day 2
Drug: Vincristine — 1,4 mg/m2 (max 2 mg) day 2
Drug: Prednisone — 40 mg/m2 day 2-6
Drug: Doxorubicin — 50 mg/m2 day 2

SUMMARY:
This is a multicenter study phase II, open-label for cardiopathic patients affected by Non-Hodgkin's lymphoma diffuse large B cell CD20 + grade IIIb follicular. The purpose is to study the feasibility of R-COMP in this cohort of patients.

ELIGIBILITY:
Inclusion Criteria:

* NHL histological diagnosis of diffuse large B cell CD20 + (de novo or shift from low-grade NHL if not pretreated), grade IIIb follicular NHL;
* Age >= 18 years;
* Presence of at least 1 factor that defines the cardiopathy;
* Life expectancy > 3 months;
* In the case of women of childbearing age absence of pregnancy at the beginning of the chemotherapy;
* Written informed consent.

Exclusion Criteria:

* Histology different from NHL diffuse large cell CD20 + or follicular IIIb
* Age < 18 years
* Inability to sign informed consent;
* HIV positivity;
* Patients HBsAg positive;
* AST/ALT > 2 times the standard;
* Bilirubin > 2 times the standard;
* Creatinine > 2.5 mg / dl;
* Location of CNS disease;
* Pregnancy ongoing;
* Damage to that organ or medical problems that could interfere with the therapy;
* Current uncontrolled infection;
* Senile dementia

Min Age: 18 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2010-05; Primary Completion 2011-05 (Actual); Study Completion 2012-05 (Estimated)

PRIMARY OUTCOMES:
Feasibility of R-COMP in cardiopathic patients | 2 years

SECONDARY OUTCOMES:
Response rates | 1 year
Progression free survival | 2 years
Overall Survival | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Michele Spina, MD, Study Director — Centro di riferimento Oncologico di Aviano
Locations (32):
- Italy (32):
  - Ospedale SS Antonio Biagio e Cesare Arrigo, Alessandria
  - Università di Bari, Bari
  - Ospedale degli Infermi, Biella
  - Spedali Civili, Brescia
  - Ospedale Civitanova Marche, Civitanova Marche
  - AO Annunziata, Cosenza
  - Ospedale San Carlo, Cosenza
  - Ospedale Vito Fazzi, Lecce
  - Istituto Scientifico Romagnolo per lo studio e la cura dei tumori (IRST), Meldola (FC)
  - A O Papardo, Messina
  - Ospedale Niguarda Cà Granda, Milan
  - Ospedale San Raffaele, Milan
  - Centro oncologico modenese, Modena
  - AO Universitaria Paolo Giaccone, Palermo
  - Ospedale La Maddalena, Palermo
  - A O Universitaria di Parma, Parma
  - Ospedale Santa Maria della Misericordia, Perugia
  - Ausl Ravenna, Ravenna
  - Ospedale Bianchi Melacrino Morelli, Reggio Calabria
  - AO Santa Maria Nuova, Reggio Emilia
  - Ausl Rimini, Rimini
  - Istituto Regina Elena, Roma
  - Ospedale Sant'Eugenio, Roma
  - Università La Sapienza, Roma
  - Clinica Humanitas, Rozzano (MI)
  - Casa sollievo della sofferenza, San Giovanni Rotondo
  - Università di Sassari, Sassari
  - Azienda Ospedaliera senese, Siena
  - Ospedale San Giovanni Battista Molinette, Torino
  - Ospedale Riuniti, Trieste
  - Santa Maria della Misericordia, Udine
  - Ospedale di circolo e Fondazione Macchi, Varese